CLINICAL TRIAL: NCT01689246
Title: Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, 15-Month Trial of TRx0237 in Subjects With Mild to Moderate Alzheimer's Disease
Brief Title: Safety and Efficacy Study Evaluating TRx0237 in Subjects With Mild to Moderate Alzheimer's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: TauRx Therapeutics Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TRx-237-015
Record Dates: First submitted 2012-09-14; First posted 2012-09-21 (Estimated); Last update posted 2018-03-14 (Actual); Status verified 2018-03

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's Disease; Alzheimer Disease; TRx0237; AD; Neurodegenerative Diseases; Dementia; Brain Diseases
MeSH Terms: conditions — Alzheimer Disease; Neurodegenerative Diseases; Dementia; Brain Diseases | interventions — hydromethylthionine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- TRx0237 250 mg/day (Experimental)
  Interventions: Drug: TRx0237 250 mg/day
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- TRx0237 150 mg/day (Experimental)
  Interventions: Drug: TRx0237 150 mg/day

INTERVENTIONS:
Drug: TRx0237 150 mg/day — TRx0237 75 mg tablets will be administered twice daily.
  Arms: TRx0237 150 mg/day
Drug: TRx0237 250 mg/day — TRx0237 125 mg tablets will be administered twice daily.
  Arms: TRx0237 250 mg/day
Drug: Placebo — Placebo tablets will be administered twice daily. The active placebo tablets include 4 mg of TRx0237 as a urinary and fecal colorant to maintain blinding; hence the placebo group will receive a total of 8 mg/day of TRx0237.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the safety and efficacy of TRx0237 in the treatment of subjects with mild to moderate Alzheimer's Disease.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of all cause dementia and probable Alzheimer's disease
* Clinical Dementia Rating (CDR) total score of 1 (mild) to 2 (moderate) and MMSE score of 14-26 (inclusive)
* Age < 90 years
* Modified Hachinski ischemic score of ≤ 4
* Females, if of child-bearing potential, must practice true abstinence or be competent to use adequate contraception and agree to maintain this throughout the study
* Subject, and/or, in the case of reduced decision-making capacity, legally acceptable representative(s) consistent with national law is/are able to read, understand, and provide written informed consent
* Has one (or more) identified adult caregiver who is willing to provide written informed consent for his/her own participation; is able to read, understand, and speak the designated language at the study site; either lives with the subject or sees the subject for ≥2 hours/day ≥3 days/week; agrees to accompany the subject to each study visit; and is able to verify daily compliance with study drug
* If currently taking an acetylcholinesterase inhibitor and/or memantine at the time of Screening, the subject must have been taking such medication(s) for ≥3 months. The dosage regimen must have remained stable for ≥6 weeks and it must be planned to remain stable throughout participation in the study.
* Able to comply with the study procedures

Exclusion Criteria:

* Significant central nervous system (CNS) disorder other than Alzheimer's disease
* Significant focal or vascular intracranial pathology seen on brain MRI scan
* Clinical evidence or history of stroke, transient ischemic attack, significant head injury or other unexplained or recurrent loss of consciousness ≥15 minutes
* Epilepsy
* Major depressive disorder, schizophrenia, or other psychotic disorders, bipolar disorder, or substance (including alcohol) related disorders
* Metal implants in the head (except dental), pacemaker, cochlear implants, or any other non-removable items that are contraindications to MRI
* Resides in hospital or moderate to high dependency continuous care facility
* History of swallowing difficulties
* Pregnant or breastfeeding
* Glucose-6-phosphate dehydrogenase deficiency
* History of significant hematological abnormality or current acute or chronic clinically significant abnormality
* Abnormal serum chemistry laboratory value at Screening deemed to be clinically relevant by the investigator
* Clinically significant cardiovascular disease or abnormal assessments
* Preexisting or current signs or symptoms of respiratory failure
* Concurrent acute or chronic clinically significant immunologic, hepatic, or endocrine disease (not adequately treated) and/or other unstable or major disease other than Alzheimer's disease
* Diagnosis of cancer within the past 2 years prior to Baseline (other than basal cell or squamous cell skin cancer or Stage 1 prostate cancer) unless treatment has resulted in complete freedom from disease for at least 2 years
* Prior intolerance or hypersensitivity to methylthioninium-containing drug, similar organic dyes, or any of the excipients
* Treatment currently or within 3 months before Baseline with any of the following medications:

  * Tacrine
  * Clozapine, olanzapine (and there is no intent to initiate therapy during the course of the study)
  * Carbamazepine, primidone
  * Drugs with a warning or precaution in the labeling about methemoglobinemia at approved doses
* Current or prior participation in a clinical trial as follows:

  * Clinical trial of a product for cognition within 3 months of Screening (unless confirmed to have been randomized to placebo)
  * A clinical trial of a drug, biologic, therapeutic device, or medical food in which the last dose/administration was received within 28 days prior to Baseline

Max Age: 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 891 (Actual)
Dates: Start 2013-01; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Change from Baseline on Alzheimer's Disease Cooperative Study - Activities of Daily Living (ADCS-ADL23) | 65 weeks
Change from Baseline on Alzheimer's Disease Assessment Scale - Cognitive Subscale (ADAS-cog11) | 65 weeks
Number of study participants who tolerate oral doses of TRx0237 as determined by safety parameter changes | 65 weeks
  Safety parameters include adverse events, vital signs, methemoglobin and oxygen saturation, physical and neurological examinations, laboratory tests (hematology, serum chemistry, and urinalysis), electrocardiograms, potential for suicide and self-harm, brain magnetic resonance imaging (MRI), and potential for serotonin toxicity

SECONDARY OUTCOMES:
Change from Baseline on Alzheimer's Disease Cooperative Study - Clinical Global Impression of Change (ADCS-CGIC) | 65 weeks
Change from Baseline on Mini-Mental Status Examination (MMSE) | 65 weeks
Change in expected decline of whole brain volume as measured by brain MRI | 39 weeks and 65 weeks

OTHER OUTCOMES:
Reduction in glucose uptake decline in the temporal lobe on 18F-fluorodeoxyglucose positron emission tomography (FDG-PET) imaging | 39 weeks and 65 weeks
Change in expected increase in ventricular volume and decline in hippocampal volume as evaluated by MRI | 39 weeks and 65 weeks
Change in resource utilization using the Resource Utilization in Dementia (RUD) Lite | 65 weeks
Change from Baseline on cerebrospinal fluid biomarkers of Alzheimer's Disease in subjects who separately consent to lumbar puncture | 65 weeks
Compare the influence of Apolipoprotein E genotype on the primary and selected secondary outcomes in subjects by or for whom legally acceptable consent is separately provided | 65 weeks

CONTACTS AND LOCATIONS:
Locations (121):
- United States (26):
  - Xenoscience, Inc/ 21st Century Neurology, Phoenix, Arizona
  - Feldman, Robert MD, Laguna Hills, California
  - University of Southern California, Los Angeles, California
  - Shankle Clinic and Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Pacific Research Network, San Diego, California
  - San Francisco Clinical Research Center, San Francisco, California
  - Yale University School of Medicine, New Haven, Connecticut
  - JEM Research, Atlantis, Florida
  - Brain Matters Research, Delray Beach, Florida
  - CNS Healthcare, Inc, Jacksonville, Florida
  - Compass Research, LLC-North Clinic, Leesburg, Florida
  - Miami Research Associates, Miami, Florida
  - Compass Research, LLC, Orlando, Florida
  - iResearch Atlanta, Decatur, Georgia
  - Alexian Brothers Neurosciences Institute, Elk Grove, Illinois
  - ActivMed Practices & Research, Methuen, Massachusetts
  - Olive Branch Family Medical, Olive Branch, Mississippi
  - Memory Enhancement Centers of America, Inc, Eatontown, New Jersey
  - CRI Worldwide, Marlton, New Jersey
  - The Cognitive Research Center of New Jersey, Springfield, New Jersey
  - Advanced Memory Research Institute of NJ PC, Toms River, New Jersey
  - Neurological Associates of Albany, P. C., Albany, New York
  - SPRI, Brooklyn, New York
  - Neurobehavioral Clinical Research, Canton, Ohio
  - The Clinical Trial Center, LLC, Jenkintown, Pennsylvania
  - FutureSearch Trials of Neurology, Austin, Texas
- Australia (9):
  - Division of Rehabilitation and Aged Care, Hornsby, New South Wales
  - Southern Neurology Pty Limited, Kogarah, New South Wales
  - Academic Department for Old Age Psychiatry, Prince of Wales Hospital, Randwick, New South Wales
  - Discipline of Psychiatry, University of Qld, Herston, Queensland
  - Royal Adelaide Hospital Memory Trials Centre, Adelaide, South Australia
  - Memory Unit, Neurology, The Queen Elizabeth Hospital, Woodville South, South Australia
  - Medical and Cognitive Research Unit, Austin Health Heidelberg Repatriation Hospital, Heidelberg West, Victoria
  - McCusker Alzheimer's Research Foundation Inc, Nedlands, Western Australia
  - Neurodegenerative Disorders Research Pty Ltd, Perth, Western Australia
- Bulgaria (2):
  - UMHAT "Alexandrovska" Clinic of Neurology Diseases Department of Neurodegenerative and Immune and Infectious Diseases of Central Nervous System with Sector for Treatment of Neuroinfections, Sofia
  - UMHAT "Alexandrovska" Clinic of Psychiatry First Department of Psychiatry, Sofia
- Canada (3):
  - Okanagan Clinical Trials, Kelowna, British Columbia
  - True North Clinical Research Kentville Inc, Kentville, Nova Scotia
  - Toronto Memory Program, North York, Ontario
- Croatia (2):
  - University Hospital Centre Zagreb, Zagreb
  - University Psychiatric Hospital Vrapce, Zagreb
- Germany (3):
  - Neurozentrum Achim Dr. med. Andreas Mahler, Achim
  - Charité, University Medicine Berlin, CBF, Neurology, Berlin
  - Memory Clinic, ECRC, Berlin
- Italy (9):
  - Neurologia Ospedale Maggiore Policlinico, Milan
  - Istituto Neurologico Carlo Besta, Milan
  - IRCCS Istituto neurologico Casimiro Mondino, Pavia
  - Clinica Neurologica, Università di Perugia-Ospedale S. Maria della Misericordia, Perugia
  - Universita' Cattolica del Sacro Cuore, Roma
  - Azienda Ospedaliera Universitaria Sant'Andrea di Roma- Unita' di Neurologia, Roma
  - Dipartimento di Neuroscienze Universita' di Torino, Torino
  - Azienda Ospedaliera S.maria Della Misericordia, Udine
  - U.O. Di Neurologia Ospedale di Circolo e Fondazione Macchi, Varese
- Malaysia (4):
  - University Kuala Lumpur Royal College of Medicine, Ipoh
  - Hospital Sultan Ismail, Johor Bahru
  - University Malaya Medical Centre, Kuala Lumpur
  - Taiping Hospital, Taiping
- Poland (9):
  - Podlaskie Centrum Psychogeriatrii, Bialystok
  - Pallmed sp zoo prowadząca NZOZ Dom Sue Ryder; Centrum Psychoneurologii Wieku Podeszłego, Bydgoszcz
  - NZOZ Wielospecjalistyczna Poradnia Lekarska SYNAPSIS, Katowice
  - Gabinet Neurologiczny, Indywidualna Specjalistyczna Praktyka Lekarska, Mosina
  - NZOZ Neuro-Kard Ilkowski i Partnerzy Spółka Partnerska Lekarzy, Poznan
  - Euromedis Sp. z o.o., Szczecin
  - Usługi Lekarskie Sp.c Palasik, Żabierek, Warsaw
  - mMED, Warsaw
  - MTZ Clinical Research Sp. z o.o., Warsaw
- Romania (8):
  - County Emergency Clinical Hospital Arad, Psychiatry Department, Arad
  - CMDTA "Neomed", Brasov
  - University Emergency Central Military Hospital "Dr.Carol Davila", Psychiatry Department, Bucharest
  - Psychomedical Consult, Bucharest
  - Clinical Municipal Hospital "Dr. Gavril Curteanu", Psychiatry Department, Oradea
  - Psychiatry Hospital "Dr. Gheorghe Preda", Center of Mental Health, Sibiu
  - Psychiatry Hospital "Dr. Gheorghe Preda", Department of Psychiatry III, Sibiu
  - Emergency Clinical County Hospital Sibiu, Neurology Department, Sibiu
- Russia (8):
  - Non-governmental Healthcare Institution "Central Clinical Hospital #6 of the JSC "Russian Railways", Moscow
  - Mental Health Research Center of the Russian Academy of Medical Sciences, Gerontopsychiatry department, Moscow
  - Mental Health Research Center of the Russian Academy of Medical Sciences, Moscow
  - CityClinical Hospital #34, City Scientific Practical Neurological Center, Novosibirsk
  - City Geriatric Medical and Social Center, Saint Petersburg
  - Saint Nicholas Psychiatric Hospital, Saint Petersburg
  - Saint Petersburg Psychoneurological Research Institute n. a. V.M. Bekhterev, Saint Petersburg
  - State Budgetary Healthcare Institution of Sverdlovsk region "Sverdlovsk Regional Clinical Psychiatric Hospital", Yekaterinburg
- Singapore (4):
  - National University Hospital (NUH), Singapore
  - National Neuroscience Institute (NNI), Singapore
  - Tan Tock Seng Hospital (TTSH), Singapore
  - Changi General Hospital, Singapore
- South Korea (10):
  - Dong-A Medical Center, Busan
  - Inha University Hospital, Incheon
  - Gachon University Gil Medical Center, Incheon
  - Seoul National University Bundang Hospital, Seongnam-si
  - Seoul National University Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Asan Medical Center, Seoul
  - Inje University Sanggye Paik Hospital, Seoul
  - Konkuk University Medical Center, Seoul
  - Seoul National University Boramae Medical Center, Seoul
- Spain (4):
  - Hospital Universitario de Ceuta, Ceuta
  - Hospital Reina Sofía, Córdoba
  - Hospital Clinico San Carlos, Madrid
  - Hospital Viamed Montecanal, Zaragoza
- Taiwan (7):
  - Changhua Christian Hospital, Changhua
  - Chang Gung Memorial Hospital, Kaohsiung, Kaohsiung City
  - China Medical University Hospital, Taichung
  - En Chu Kong Hospital, Taipei
  - National Taiwan University Hospital, Taipei
  - National Yang-Ming University School of Medicine, Taipei
  - Chang Gung Memorial Hospital, Linkou, Taoyuan District
- United Kingdom (13):
  - NHS Grampian, Department of Old Age Psychiatry Royal Cornhill Hospital, Aberdeen
  - RICE - The Research Institute for the Care of Older People, Bath
  - Belfast Health and Social Care Trust (BHSCT), Belfast
  - The Barberry Centre, Birmingham
  - MAC Clinical Research Ltd, Blackpool
  - MAC Clinical Research Ltd, Bradford
  - MAC Clinical Research Ltd, Cannock
  - MAC Clinical Research Ltd, Leeds
  - Re: Cognition Health Ltd., London
  - Charing Cross Hospital, London
  - Dementia Research Centre, London
  - MAC Clinical Research Ltd, Manchester
  - Southampton General Hospital, Southampton

REFERENCES:
- [Derived] Gauthier S, Feldman HH, Schneider LS, Wilcock GK, Frisoni GB, Hardlund JH, Moebius HJ, Bentham P, Kook KA, Wischik DJ, Schelter BO, Davis CS, Staff RT, Bracoud L, Shamsi K, Storey JM, Harrington CR, Wischik CM. Efficacy and safety of tau-aggregation inhibitor therapy in patients with mild or moderate Alzheimer's disease: a randomised, controlled, double-blind, parallel-arm, phase 3 trial. Lancet. 2016 Dec 10;388(10062):2873-2884. doi: 10.1016/S0140-6736(16)31275-2. Epub 2016 Nov 16. PMID 27863809
- See also: Alzheimer's Survey — http://www.AlzheimersStudies.com